CLINICAL TRIAL: NCT06314698
Title: A Multicenter, Randomized, Controlled, Non-inferiority Study of Narlumosbart Compared With Denosumab in the Treatment of Bone Disease in Patients With Multiple Myeloma
Brief Title: Narlumosbart Compared With Denosumab in Patients With Multiple Myeloma Bone Disease
Status: Not yet recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: RenJi Hospital (Other)
Collaborators: Shanghai JMT-Bio Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: IIT-2024-0011
Record Dates: First submitted 2024-03-10; First posted 2024-03-18 (Actual); Last update posted 2024-03-18 (Actual); Status verified 2024-03

CONDITIONS: Multiple Myeloma; Bone Diseases
MeSH Terms: conditions — Multiple Myeloma; Bone Diseases | interventions — Denosumab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Narlumosbart (Experimental): 120 mg SC Q4W, up to 2 years.
  Interventions: Drug: Narlumosbart
- Denosumab (Active Comparator): 120 mg SC Q4W, up to 2 years.
  Interventions: Drug: Denosumab

INTERVENTIONS:
Drug: Narlumosbart — Administered by subcutaneous injection once every 4 weeks.
  Other Names: Narlumosbart Injection, JMT103
  Arms: Narlumosbart
Drug: Denosumab — Administered by subcutaneous injection once every 4 weeks.
  Other Names: XGEVA®, AMG 162
  Arms: Denosumab

SUMMARY:
The purpose of this study is to determine if narlumosbart is non-inferior to denosumab in the treatment of bone diseases from multiple myeloma (MM).

DETAILED DESCRIPTION:
Multiple myeloma is a plasma cell dyscrasia with a high likelihood of causing bone disease (ie, multiple myeloma-related bone disease); as a result, up to 80% of patients with newly diagnosed multiple myeloma present with osteolytic lesions.

Denosumab is recommended for the treatment of newly diagnosed multiple myeloma, and for patients with relapsed or refractory multiple myeloma with evidence of multiple myeloma-related bone disease.

Narlumosbart is a recombinant, fully human, anti-receptor activator of nuclear factor kappa-Β ligand (RANKL) IgG4 monoclonal antibody. Changing the IgG2 Fc portion of denosumab to IgG4, results in increased stability, higher specificity and affinity for RANKL than denosumab. The objective of this phase III trial is to compare the efficacy and safety between Narlumosbart and denosumab in patients with bone diseases from newly diagnosed multiple myeloma.

ELIGIBILITY:
Inclusion Criteria:

1. Subjects fully understand and voluntarily participate in this study and sign the informed consent;
2. Age≥18, no gender limitation;
3. Active multiple myeloma patients with newly diagnosed by International Myeloma Working Group (IMWG) 2014 criteria;
4. Measurable lesion per at least one of the following criteria : Serum monoclonal protein ≥10 g/L; Urinary monoclonal protein ≥200 mg/24h; Serum free Light Chain (FLC) assay showed an involved FLC level ≥100 mg/L with abnormal ratio for FLC (κ/λ);
5. Radiographic [X-ray, computer tomography (CT), magnetic resonance imaging (MRI), positons emission tomography coupled with a computer tomography (PET-CT)] evidence of at least one lytic bone lesion;
6. Plan to receive primary frontline anti-myeloma therapies, or receiving less than one cycle of frontline anti-myeloma therapy (less than 30 days, does not include radiotherapy or a single short course of steroid), the treatment regimens were limited to VRd, D-VRd, DRd, and VCd;
7. Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1, or 2
8. Adequate organ function, as defined by the following criteria (per laboratory values):

   1. Liver function: Serum total bilirubin ≤ 2.0 x upper limit of normal (ULN), Serum alanine aminotransferase ≤ (ALT) 2.0 x ULN, Serum aspartate aminotransferase (AST) ≤ 2.0 x ULN
   2. Renal function: Serum creatinine clearance (CrCL) ≥ 30 mL/min, calculated by the Cockcroft-Gault formula
   3. Serum calcium or albumin-adjusted serum calcium ≥2.0 mmol/L (8.0 mg/dL) and ≤ 2.9 mmol/L (11.5 mg/dL)
9. Reproductive potential subjects should be receiving effective contraception (Both male and female reproductive potential subjects, from the date of signing the informed consent to 6 months after the end of treatment);
10. Expected survival time ≥ 3 months;

Exclusion Criteria:

1. POEMS syndrome;
2. Plasma cell leukemia;
3. Prior history or current evidence of osteonecrosis/osteomyelitis of the jaw; Non-healed dental/oral surgery, including tooth extraction; Active dental or jaw condition which requires oral surgery; Planned invasive dental procedures;
4. Planned radiation therapy or Orthopedic surgery;
5. Prior administration of denosumab or bisphosphonates;
6. Patients with active bone metabolic diseases (Paget disease of bone, Cushing syndrome and hyperprolactinemia), rheumatoid arthritis, uncontrolled hyper/hypothyroidism or hyper/hypoparathyroidism;
7. Uncontrolled concurrent diseases, including but not limited to: symptomatic congestive heart failure, hypertension (blood pressure remains > 150/90 mmHg after standard therapy), unstable angina, arrhythmia requiring medication or instruments, history of myocardial infarction within 6 months, echocardiography showing left ventricular ejection fraction <50%;
8. Active bacterial or fungal infections requiring systemic treatment within 7 days before randomization;
9. Known infection with human immunodeficiency virus (HIV), active infection with Hepatitis B virus (positive hepatitis B surface antigen and positive HBV-DNA) or Hepatitis C virus(positive hepatitis C surface antigen and positive HCV-RNA);
10. Pregnancy (serum β-HCG positive) or lactation;
11. Use of any of the following anti-bone metabolism drugs within 6 months before enrollment:

    1. parathyroid hormonerelated peptides
    2. calcitonin
    3. osteoprotegerin
    4. mithramycin
    5. strontium ranelate
12. Known sensitivity to narlumosbart, denosumab, calcium or vitamin D;
13. Any other factors not suitable for participation in this study that in the opinion of the investigator.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 478 (Estimated)
Dates: Start 2024-04-01 (Estimated); Primary Completion 2024-12-31 (Estimated); Study Completion 2027-04-30 (Estimated)

PRIMARY OUTCOMES:
Percent change from baseline in urinary N-terminal telopeptide of type 1 collagen corrected for urinary creatinine (uNTx/uCr) at week 13 | From baseline to week 13
  Compare narlumosbart and denosumab for percentage change in bone turnover marker (BTM) - urinary N-terminal telopeptide of type 1 collagen (uNTx) corrected for urinary creatinine (uCr) (uNTx/uCr from baseline to week 13)

SECONDARY OUTCOMES:
The proportion of subjects with a change in uNTx/uCr greater than 65% from baseline to week 13 | From baseline to week 13
  Compare narlumosbart and denosumab for the proportion of subjects with a change in uNTx/uCr greater than 65% from baseline to week 13 (uNTx/uCr from baseline to week 13 >65%)
Time to first on-study skeletal related event | From baseline to 90 days after the last dose, up to approximately 30 months
  A skeletal-related event (SRE) is defined as one of the following: pathologic fracture, radiation therapy to bone, surgery to bone, or spinal cord compression. Time to first on-study SRE is defined as the time interval (in days) from the randomization date to the date of first occurrence of on-study SRE
Percentage of participants with an on-study SRE at different time points | Months 3, 6, 12, 18 and 24
  A skeletal-related event (SRE) is defined as one of the following: pathologic fracture, radiation therapy to bone, surgery to bone, or spinal cord compression.
  Percentage of participants with an on-study SRE at 3, 6, 12, 18 and 24 months
Time to first and subsequent on-study SRE | From baseline to 90 days after the last dose, up to approximately 30 months
  Time to first on-study SRE is defined as the time interval (in days) from the randomization date to the date of first occurrence of on-study SRE.
  Time to a subsequent SRE is defined, similarly to the time to first on-study SRE, as the time interval from the randomization date to the date of a subsequent occurrence of on-study SRE, which had to be at least 21 days after the previous SRE.
Percent changes of serum bone alkaline phosphatase (BALP) and serum C-terminal telopeptide of type 1 collagen (sCTX-I) | From baseline to week 13
  Compare the changes of BALP and sCTX-I from baseline to weeks 13
Overall Survival | From baseline to 90 days after the last dose, up to approximately 30 months
  Overall survival was defined as the time interval (in days) from the randomization date to the date of death.
Incidence and type of adverse events (AEs) | From the first dose finished to 28 days after the last dose
  To identify the incidence and the type of AEs, including abnormalities in clinical, laboratory assessments, ECGs, echocardiography, vital sign assessments, and physical exams.

CONTACTS AND LOCATIONS:
Overall Officials: Jian Hou, M.D., Principal Investigator — RenJi Hospital

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Dhillon S. Narlumosbart: First Approval. Drugs. 2024 Jan;84(1):105-109. doi: 10.1007/s40265-023-01985-3. PMID 38112898